CLINICAL TRIAL: NCT00359463
Title: An Open-Label, Non-Randomized Pharmacokinetic and Safety Study of a Single Oral Dose of 50mg Eltrombopag in Healthy Subjects and in Volunteers With Mild, Moderate or Severe Hepatic Impairment
Brief Title: Study Of Eltrombopag in Healthy Subjects and Volunteers With Mild, Moderate or Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRA103452
Record Dates: First submitted 2006-07-28; First posted 2006-08-02 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: hepatitis C-associated thrombocytopenia; chemotherapy induced thrombocytopenia; thrombocytopenia; hepatic impairment; chronic immune thrombocytopenia purpura
MeSH Terms: conditions — Purpura; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Active Comparator): Subjects will receive a single 50 mg oral dose of eltrombopag.
  Interventions: Drug: eltrombopag
- Subjects with hepatic impairment (Experimental): Subjects with mild, moderate or severe hepatic impairment will receive a single 50 mg oral dose of eltrombopag.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — Subjects will be administered a single oral dose of 50 mg eltrombopag.

SUMMARY:
The main purpose of this study is to compare how one 50mg tablet of SB-497115 is broken down in the body by healthy subjects versus subjects with mild, moderate or severe liver problems. The study is also being done to 1) check on how well the study drug is tolerated by healthy subjects versus those with liver problems and 2) to check if liver impairment affects how the study drug binds to protein in the blood.

ELIGIBILITY:
Inclusion criteria:

* Healthy or have liver impairment
* Females(the following requirement applies only if able to have children): agree to doctor approved birth control methods, or partner has had a vasectomy.
* Body mass index (BMI-within acceptable range)
* Negative drug, alcohol, and HIV tests

Exclusion criteria:

* Taking a medication or therapy not approved by the study doctor
* Rapidly changing liver function
* Kidneys not working well
* Drug or alcohol abuse within past 6 months
* Used an investigational drug in the past 30 days
* Females that are pregnant or nursing
* Have active hepatitis B or C
* History of blood disorders
* History of various heart conditions (as noted by study doctor)
* Blood clotting problems or blood abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-04-18 (Actual); Primary Completion 2007-03-07 (Actual); Study Completion 2007-03-07 (Actual)

PRIMARY OUTCOMES:
Plasma levels and protein binding of eltrombopag | Day 1 to Day 6

SECONDARY OUTCOMES:
Safety will be monitored by: - clinical lab tests - vital signs - electrocardiograms - monitoring for adverse events - physical exams - eye exams | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Orlando, Florida
- Australia (2):
  - GSK Investigational Site, Randwick, Sydney, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
- GSK Investigational Site, Christchurch, New Zealand

REFERENCES:
- [Background] Bauman JW, Vincent CT, Peng B, Wire MB, Williams DD, Park JW. Effect of hepatic or renal impairment on eltrombopag pharmacokinetics. J Clin Pharmacol. 2011 May;51(5):739-50. doi: 10.1177/0091270010372106. Epub 2010 Jul 27. PMID 20663991
- See also: Results for study 103452 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/TRA103452?search=study&search_terms=103452#rs